CLINICAL TRIAL: NCT01269398
Title: Achieving Solide Fusion, Comibing the GO-LIF Procedure for Spinal Fixation and Stabilization With Percutaneous Posetrior Facets Fusion.
Brief Title: GO-LIF With Percutaneous Facet Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Yair Barzilay, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group
Other Study IDs: BARZ-004-HMO-CTIL
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Lumbar Fusion

ARMS (2):
- GO-LIF procedure, posetrior facets fusion (No Intervention)
- solid fusion, GO-LIF procedure (Other): ability to achieve solid fusion, comibing the GO-LIF procedure for spinal fixation and stabilization with percutaneous posetrior facets fusion
  Interventions: Device: GO-LIF and SpineAssist SYSTEMS

INTERVENTIONS:
Device: GO-LIF and SpineAssist SYSTEMS
  Arms: solid fusion, GO-LIF procedure

SUMMARY:
Utilization of trans-pedicular trans-discal implants for stabilization of a single lumbar motion segment, in conjunction with posterior facets fusion. The trajectories are planned and achieved by means of the SpineAssist® system - a computerized, image-based guidance system that assists surgeons in precisely guiding spinal surgical tools and implants in line with a CT-based pre-operative plan. GO-LIF and SpineAssist are CE marked products.

Thy study's objective is to to collect data regarding the ability to achieve solide fusion, comibing the GO-LIF procedure for spinal fixation and stabilization with percutaneous posterior facets fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally-mature patients requiring single-level instrumented fusion from L1 to S1
2. Men and women, 18-80 years of age.
3. Unequivocal medical indication for the fixation surgery of a single motion segment of the lumbar spine.
4. Correct coronal profile of the lumbar spine. An asymmetric collapse of the disk space in the coronal plane between the vertebral bodies envisioned for instrumentation is by itself not an exclusion criterion.
5. Patient may have, but is not required to, secondary diagnosis of any one of the following:

   * Degenerative spondylolisthesis (Grades 1 and 2) in the sagittal plane with preserved or normal sagittal alignment
   * Spinal stenosis (Not excluding patient with a need to decompression )
6. ODI cut-off for inclusion, lower than or equal to 40 for ODI
7. VAS cut-off for inclusion, lower than or equal to 9
8. Patient is willing and able to comply with study requirements, including follow-up schedule and postoperative management program
9. Patient must understand and sign informed consent

Exclusion Criteria:

1. Lumbar hyperlordosis > 70° between the end plate of the lumbar vertebral body 1 and the end plate of the sacral vertebral body 1.
2. Deformities of the vertebral bodies envisioned for instrumentation or the sacrum.
3. Spondylolisthesis > grade 2 acc. to Meyerding.
4. Scoliosis and other deformities in the coronal plane.
5. Fractures of the vertebrae envisioned for instrumentation.
6. Osteoporosis or osteopenia (see below for examination criteria).
7. Therapy with systemic corticosteroids or immunosuppressants.
8. Bone metabolism diseases, such as osteomalacia or Paget's disease.
9. Post inflammatory instability of the vertebral spine.
10. State after radiation therapy of the relevant vertebral spine region.
11. Current Marcoumar or heparin therapy for more than 6 months at the time of operation.
12. Malignant diseases with or without bone metastases.
13. Immunologic-inflammatory diseases (e.g., rheumatoid arthritis).
14. Diabetes mellitus.
15. Infectious diseases.
16. More than one motion segments requiring treatment.
17. Prior percutaneous vertebral augmentation procedure (e.g., vertebroplasty, kyphoplasty) at index or adjacent level.
18. Prior fusion attempts at the involved levels.
19. Clinically or radiographically compromised vertebral bodies at the superior vertebra of the affected level or compromised pedicles at the inferior vertebra of the affected level due to current or past trauma such that a Onyx Spinal System can not be implanted
20. Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least 5 years.
21. Coagulopathy or inability to reverse anti-coagulant therapy (both during and approximately 24 hours post-procedure).
22. Metabolic bone disease such as Paget's disease, osteopenia or osteomalacia.
23. Severe diabetes mellitus requiring daily insulin management.
24. Haemorrhagic diasthesis.
25. Coagulation disorders, or severe cardiopulmonary disease.
26. Active systemic infection (including AIDS, HIV and Hepatitis) or active infection at surgical site.
27. Rheumatoid arthritis or other autoimmune disease.
28. Morbid obesity, defined as having a Body Mass Index of 40 or higher or more than 100 pounds over weight.
29. Conditions or medications that may interfere with bony/soft tissue healing (e.g., long term steroid use).
30. Any medical condition that would preclude the patient from having surgery, impede the benefit of spinal implant surgery or impede the patient from completing the post operative rehabilitation plan.
31. Pregnancy, current or planned during the duration of the study.
32. Subject has a history of substance abuse (e.g., recreational drugs, narcotics, or alcohol) within the last 12 months.
33. Known allergy to titanium or titanium alloys.
34. Bone growth stimulator use anywhere in the body within the last 30 days.
35. In active spinal litigation.
36. Degenerative spondylolisthesis (Grades 3 and above)
37. Is currently involved in a study of another investigational product for similar purpose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
percutaneous posetrior facets fusion | 1 year
  Fusion will be determined by and evaluated by the acheivement of a fusion and controled after 1 year by a CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel